CLINICAL TRIAL: NCT01071200
Title: A Phase III, Multicentric, Randomized, Open, Comparative Study to Evaluate if the Addition of Recombinant Human Luteinising Hormone [r-hLH (Luveris®)] to Follicle Stimulating Hormone (FSH) From Day 8 of Ovarian Stimulation is Able to Decrease Total FSH Dose and to Improve Cycle Outcome in Infertile Women Undergoing Assisted Reproduction Technology (ART), Who Required High FSH Dose in a Previous Cycle
Brief Title: Study to Evaluate if the Addition of r-hLH (Luveris®) to FSH From Day 8 of Ovarian Stimulation is Able to Decrease Total FSH Dose and to Improve Cycle Outcome in Infertile Women Undergoing ART, Who Required High FSH Dose in a Previous Cycle
Acronym: Luveris in ART
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.P.A., Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMP25289; 2004-002218-13 (EudraCT Number); NCT00267761 (obsolete NCT alias)
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Reproductive Techniques, Assisted
Keywords: Reproductive Techniques, Assisted; Recombinant human follicle stimulating hormone (r-hFSH); Recombinant leutinizing hormone (r-hLH)
MeSH Terms: conditions — Helping Behavior

ARMS (2):
- A (Experimental): Subjects treated with r-hFSH and r-hLH (2:1 ratio of r-hFSH:r-hLH)
  Interventions: Drug: Recombinant human Follicle Stimulating Hormone (r-hFSH) and Recombinant human Luteinizing Hormone (r-hLH)
- B (Active Comparator): Subjects treated with r-hFSH alone
  Interventions: Drug: r-hFSH

INTERVENTIONS:
Drug: Recombinant human Follicle Stimulating Hormone (r-hFSH) and Recombinant human Luteinizing Hormone (r-hLH) — One r-hFSH and one r-hLH injection subcutaneously (s.c.) once daily during the treatment phase from Day 8 of stimulation until injection of human chorionic gonadotropin (hCG) or cancellation of the treatment cycle.
  Other Names: r-hLH; r-hFSH
  Arms: A
Drug: r-hFSH — One r-hFSH injection s.c. once daily during the treatment phase from Day 8 of stimulation until injection of hCG or cancellation of the treatment cycle.
  Arms: B

SUMMARY:
The present study was designed to investigate, in hyporesponder subjects, that required in a previous assisted reproductive technologies (ART) cycle follicle stimulating hormone (FSH) >3500 International Unit (IU), the possibility to decrease through recombinant human luteinizing hormone (r-hLH) supplementation, the FSH amount per oocytes retrieved and in the mean time to improve the overall cycle outcome.

DETAILED DESCRIPTION:
Recombinant human follicle stimulating hormone (r-hFSH), which totally lacks LH activity, is widely used to induce multiple follicle development in women under pituitary desensitization, in order to submit them to treatment with assisted reproduction techniques (ART). Clinical experience from hypogonadotropic-hypogonadic women suggests that while FSH alone is sufficient to induce follicle development, LH plays a significant part in final follicle maturation, estrogen synthesis and optimal endometrium growth.

This was a phase III, multicentre, randomized, open-label comparative study to evaluate if the addition of r-hLH (Luveris) in a 2:1 ratio to FSH from day 8 of ovarian stimulation is able to decrease the total FSH dose and to improve cycle outcome in 250 infertile women undergoing ART, who required high FSH dose in a previous cycle (≥ 3500 IU). Subjects who have met all the inclusion criteria, achieved pituitary desensitization and started controlled ovarian hyperstimulation (COH) treatment with FSH, on stimulation day 8 (S8) received an identification number and will be allocated to one of the two following arms:

Arm : FSH + r-hLH (2:1 ratio of FSH:r-hLH), Arm : FSH alone. Treatment with Luveris was commenced on day 8 (S8) and continued until injection of hCG or cancellation of the treatment cycle.

Monitoring of stimulation, FSH dose escalation, criteria for injection of hCG, ovum pick up, embryo transfer and pregnancy confirmation took place according to standard management practice. The in-vitro fertilization (IVF) or intracytosolic sperm injection (ICSI) procedure, including luteal phase support, was performed according to each centres' normal procedures.

The subjects were followed up and the treatment outcome (menstruation or pregnancy) was recorded. The delivery outcome for any pregnant subjects was recorded in the Case Report Form (CRF).

Information on the delivery outcome for each pregnancy was collected. Information on adverse events was collected during the study period.

OBJECTIVES

The primary objective of the study was:

To determine whether the addition of r-hLH (Luveris) from day 8 of ovarian stimulation reduces the FSH dose needed to obtain/retrieve each oocyte.

The secondary objectives of the study were:

* To determine whether the addition of Luveris to FSH at day 8 of ovarian stimulation improves cycle outcome based on secondary endpoints
* To determine the safety of Luveris in this indication

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal infertile woman, aged 18 to 40 years inclusive, who wishes to conceive
* Regular, spontaneous menstrual cycle of 25-35 days
* Body mass index (BMI) ≤ 28
* FSH ≤ 10 IU/L (follicular phase, days 2-5)
* Prolactin (PRL) within the normal ranges
* Evidence of both ovaries by ultrasound scan
* Women undergoing IVF-Embryo Transfer (ET) or ICSI, down regulated with Gonadotropin releasing hormone analogues (GnRHa) (daily dose) under controlled ovarian hyperstimulation (COH) with FSH
* Washout > 90 days from last dose of clomiphene or gonadotrophin, before ongoing COH cycle
* Only one previous IVF-ET or ICSI cycle (in the last 9 months preceding the ongoing COH cycle) resulted in a hypo-response properly documented (from 6 to 12 oocytes with a total FSH dose ≥ 4000 IU)
* Negative pregnancy hCG test (urine or blood sample) before the ongoing COH cycles
* Willing and able to comply with the protocol for the duration of the study
* Written informed consent before applying any procedure related to the study protocol, which is not part of routine medical care, with the understanding that consent may be withdrawn by the subject at any time, without prejudice on their future medical care

Exclusion Criteria:

* Oligo/Anovulatory cycles (World Health Organization [WHO] I and II)
* Male partner azoospermia (assessed within the last 12 months)
* Follicular phase (day 2-5) FSH > 10 IU/L even if only once observed in the medical history
* Abnormal cervical cytology (assessed within the last 12 months)
* History of unexplained gynecologic hemorrhage
* Any contraindication to pregnancy
* Known allergy to gonadotrophin
* Any clinically important systemic disease (e.g. insulin-dependent diabetes mellitus, epilepsy, serious migraine, intermittent purpura, hepatic, renal or cardiovascular disease, serious corticoid-dependent asthma) which constitutes a contraindication to gonadotropin use
* Any medical condition which, according to the investigator's judgement, may affect the absorption, distribution, metabolism or excretion of the drug. In case of doubt, inclusion of the subject in question should be discussed with the Medical Responsible of Serono
* Known Human Immunodeficiency Virus (HIV) positivity
* Any substance abuse or history of drugs or alcohol abuse within the past 5 years
* Prior inclusion in the present study or simultaneous inclusion in a clinical study of another drug
* Refusal or inability to comply with the protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 133 (Actual)
Dates: Start 2005-03; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Longobardi, Study Director — Merck Serono S.P.A., Italy
Locations (1):
- Merck Serono S.p.A., Roma, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- FSH + rhLH: Follicle-stimulating hormone (FSH) injection administered according to investigator's discretion till Day 8 of stimulation period (S8) and treatment with recombinant human luteinizing hormone (rhLH, Luveris) injection 150 International Units (IU) subcutaneously (s.c.) daily was started from S8 until recombinant human choriogonadotropin (r-hCG) administration day. r-hLH was administered in a 2:1 ratio (FSH:r-hLH).
- Follicle-stimulating Hormone (FSH): FSH injection s.c. administered according to investigator's discretion till r-hCG administration day.
Period: Overall Study
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Started | 67 | 66
Completed | 60 | 63
Not Completed | 7 | 3
Not completed — Lack of ovarian response | 1 | 1
Not completed — No fertilization | 4 | 0
Not completed — No oocytes retrieved | 1 | 1
Not completed — Ovarian Hyper Stimulation Syndrome | 1 | 0
Not completed — No viable embryos | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH) | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (2.9) | 35.0 (3.8) | 35.3 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 66 | 133
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Dose of Follicular Stimulating Hormone (FSH) for Retrieved Oocytes
Time Frame: Baseline (Stimulation day 8 [S8]) until hCG day
Population: Modified intention-to-treat (mITT) population included all randomized participants who entered in the experimental phase at S8. Here "N" represents number of participants analyzed for this measure.
Measure: Mean (Standard Deviation); unit: IU
Groups:
- Follicle-stimulating Hormone (FSH): FSH injection administered according to investigator's discretion till r-hCG administration day.
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 64 | 64
IU
  Baseline (S8) | 904.6 (1068.1) | 703.3 (924.5)
  Baseline (S8) until hCG day | 388.5 (631.3) | 318.5 (534.0)

2. Secondary Outcome: Mean Total Follicle Stimulating Hormone (FSH) and Recombinant Human Luteinizing Hormone (r-hLH) Dose
Time Frame: Baseline (S8) until hCG day
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
IU
  Total FSH dose | 1434.0 (678.1) | 1595.0 (796.4)
  Total r-hLH dose | 575.9 (273.0) | 0 (0)

3. Secondary Outcome: Mean Number of Ovarian Stimulation Days
Time Frame: Baseline (S8) until hCG day
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Mean (Full Range); unit: Days
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
Days | 4.6 [2.0 to 10.0] | 4.8 [1.0 to 9.0]

4. Secondary Outcome: Change From Baseline in Oestradiol (E2) Levels at Human Choriogonadotropin (hCG) Day
Time Frame: Baseline (S8) and hCG day
Population: mITT population included all randomized participants who entered in the experimental phase at S8. Here "N" represents number of participants analyzed and "n" represents the number of participants with plasma E2 levels at specified time points for respective treatment groups.
Measure: Mean (Standard Deviation); unit: picogram/milliter (pg/mL)
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 59 | 59
picogram/milliter (pg/mL)
  Baseline (n = 59,59) | 516.1 (353.6) | 518.9 (334.2)
  Change at hCG day (n = 40,47) | 1391.6 (743.4) | 1179.9 (746.5)
Statistical Analysis 1: Comparison: FSH + rhLH vs Follicle-stimulating Hormone (FSH); Change at hCG day : Wilcoxon two sample test was used to calculate p-value; Test type: Superiority or Other; p = 0.07, Wilcoxon two sample test

5. Secondary Outcome: Mean Total Number of Retrieved Oocytes
Description: Mean number of oocytes retrieved on the day of ovum pick up (OPU) was counted. Oocyte retrieval is a technique used in in-vitro fertilization in order to remove oocytes from the ovary of the female, enabling fertilization outside the body.
Time Frame: 34-36 hours post-hCG (OPU)
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
oocytes | 7.0 (4.6) | 7.8 (3.9)

6. Secondary Outcome: Mean Number of Mature Oocytes (Metaphase II)
Description: Mean number of metaphase II oocytes was counted for participants undergoing ovum pick up for IntraCytoplasmic Sperm Injection (ICSI). ICSI is a procedure in which a single spermatozoon is injected into the oocyte cytoplasm. Metaphase II stage of the oocyte was classified as the time at which the first polar body was observed microscopically. Metaphase II oocytes are a sub-group of the total number of oocytes.
Time Frame: 34-36 hours post-hCG (OPU)
Population: mITT population included all randomized participants who entered in the experimental phase at S8. Here "N" represents those participants undergoing ICSI whose oocytes were assessed for maturity (Metaphase II) using a microscope.
Measure: Mean (Standard Deviation); unit: Metaphase II Oocytes
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 59 | 62
Metaphase II Oocytes | 5.1 (3.7) | 5.7 (3.2)

7. Secondary Outcome: Fertilization Rate
Description: Fertilization rate was measured as the ratio between number of fertilized oocytes and number of inseminated oocytes (maximum 3).
Time Frame: 12-18 day post-hCG and/or Week 7
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
ratio | 0.85 (0.29) | 0.89 (0.20)

8. Secondary Outcome: Number of Obtained Embryos
Description: Total number of obtained embryos with maximum 3 inseminated oocytes was calculated.
Time Frame: Day 3 post-hCG (Embryo transfer [ET])
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Number; unit: embryos
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
embryos | 142 | 158

9. Secondary Outcome: Number of Transferred Embryos
Description: Embryo transfer is the procedure in which one or more embryos are placed in the uterus or Fallopian tube.
Time Frame: Day 3 post-hCG (ET)
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Number; unit: embryos
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
embryos | 60 | 63

10. Secondary Outcome: Percentage of Participants With Pregnancy
Time Frame: 12-18 day post-hCG and/or Week 7
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Number; unit: percentage of participants
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
percentage of participants | 29.9 | 30.8

11. Secondary Outcome: Percentage of Participants With Clinical Pregnancy
Description: Clinical pregnancy is defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.
Time Frame: 12-18 day post-hCG and/or Week 7
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Number; unit: percentage of participants
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
percentage of participants | 23.9 | 18.5

12. Secondary Outcome: Percentage of Participants With Implantation
Description: Implantation is the attachment and subsequent penetration by the zona-free blastocyst (usually in the endometrium) that starts five to seven days after fertilization.
Time Frame: 12-18 day post-hCG and/or Week 7
Population: mITT population included all randomized participants who entered in the experimental phase at S8.
Measure: Number; unit: percentage of participants
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 65
percentage of participants | 13.38 | 11.39

13. Secondary Outcome: Number of Participants With Ovarian Hyper Stimulation Syndrome (OHSS)
Description: OHSS is an exaggerated systemic response to ovarian stimulation characterized by a wide spectrum of clinical and laboratory manifestations. It is classified as mild, moderate or severe according to the degree of abdominal distention, ovarian enlargement and respiratory, haemodynamic and metabolic complications.
Time Frame: Baseline (S8) until 12-18 day post-hCG and/or Week 7
Population: Safety population included all the randomized participants who received at least one dose of the study drug.
Measure: Number; unit: participants
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 66
participants
  Mild OHSS | 0 | 0
  Moderate OHSS | 1 | 0
  Severe OHSS | 0 | 0

14. Secondary Outcome: Number of Cycles Cancelled Due to Risk of OHSS
Description: as for outcome 13
Time Frame: Baseline (S8) until 12-18 day post-hCG and/or Week 7
Population: Safety population included all the randomized participants who received at least one dose of the study drug.
Measure: Number; unit: cycles
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Number analyzed (Participants) | 67 | 66
cycles | 1 | 0

ADVERSE EVENTS:
Time Frame: AEs are collected on an ongoing basis from day of written informed consent. All new AEs must be recorded until the post-treatment safety, on day 12-18 post-hCG administration. AEs are classified as pre-treatment, treatment-emergent and post-treatment.
Description: Pre-Treatment:Medical conditions present at the initial study visit that did not worsen in severity or frequency during the study;Treatment-Emergent: If the onset date of the AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of the AE was post-hCG Days 12 - 18 for participants who completed the study.
Arm/Group | FSH + rhLH | Follicle-stimulating Hormone (FSH)
Serious Adverse Events (participants affected / at risk) | 1/67 | 2/66
Other Adverse Events (participants affected / at risk) | 2/67 | 0/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSH + rhLH (N=67) | Follicle-stimulating Hormone (FSH) (N=66)
Left ectopic pregnancy (General disorders) | 0 | 1
Cerclage (General disorders) | 1 | 0
Renal colic (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSH + rhLH (N=67) | Follicle-stimulating Hormone (FSH) (N=66)
Ovarian Hyper Stimulation Syndrome (General disorders) | 1 | 0
Urticaria post intake of food (fish) (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other